CLINICAL TRIAL: NCT06806852
Title: A Phase Ib Open Label Randomised Clinical Trial to Evaluate Safety and Efficacy of BI 770371 in Combination With Pembrolizumab With or Without Cetuximab Compared With Pembrolizumab Monotherapy for the First-line Treatment of Patients With Metastatic or Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: A Study to Test Whether Treatment With BI 770371 in Combination With Pembrolizumab With or Without Cetuximab Helps People With Head and Neck Cancer Compared With Pembrolizumab Alone
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1501-0002; 2024-517091-38-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab
- Pembrolizumab + BI 770371 (Experimental)
  Interventions: Drug: BI 770371; Drug: Pembrolizumab
- Pembrolizumab + BI 770371 + Cetuximab (Experimental)
  Interventions: Drug: BI 770371; Drug: Pembrolizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: BI 770371 — BI 770371
  Arms: Pembrolizumab + BI 770371; Pembrolizumab + BI 770371 + Cetuximab
Drug: Pembrolizumab — Pembrolizumab
Drug: Cetuximab — Cetuximab
  Arms: Pembrolizumab + BI 770371 + Cetuximab

SUMMARY:
This study is open to adults with head and neck cancer. The purpose of this study is to find out whether combining different study medicines makes tumors shrink in people with head and neck cancer.

The tested medicines in this study are antibodies that act in different ways against cancer. BI 770371 and pembrolizumab may help the immune system fight cancer. Cetuximab blocks growth signals and may prevent the tumor from growing.

Participants are put into 3 groups randomly. Each group receives a different combination of study medicines. All study medicines are given as an infusion into a vein at the study site.

Participants can stay in the study as long as they benefit from treatment. Doctors regularly check the size of the tumor and check whether it has spread to other parts of the body. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic or recurrent HNSCC of the primary tumour location of oral cavity, oropharynx, hypopharynx, and larynx not amenable to locoregional treatment with curative intent.
* Willingness to provide pretreatment (baseline) biopsy/tissue to the sponsor (fresh or archival one). A newly obtained biopsy is preferred but an archival sample is acceptable, with tumor tissue (formalin fixed paraffin embedded [FFPE] block preferred, or at least 10 freshly sectioned unstained FFPE slides) from a core or excisional biopsy. Any deviation from this rule requires approval by the sponsor. Details on the requirements for archival tumour tissue and on biopsy sample collection are provided in the Laboratory Manual.
* Patients who have not received prior systemic treatment for metastatic or recurrent HNSCC. Systemic therapy (including cetuximab) which was completed more than 6 months prior to progression of disease if given as part of multimodal treatment for locally advanced disease is allowed.
* Patients who do not have contraindications to pembrolizumab monotherapy according to pembrolizumab local label, guidelines, treatment standards, regulations or the document (label of another country if pembrolizumab local label is not available) provided in the investigator site file (ISF) by the sponsor.
* Patients who do not have contraindications to treatment with cetuximab according to cetuximab local label, guidelines, treatment standards, regulations, or the document (label of another country if cetuximab local label is not available) provided in the ISF by the sponsor.
* Presence of at least one measurable non-central nervous system (CNS) lesion (according to RECIST v1.1.).
* Further inclusion criteria apply.

Exclusion Criteria:

* Nasopharyngeal carcinoma (NPC) of any histology, primary tumour location at nasal cavity, paranasal sinuses of any histology, any cancer of unknown primary.
* Any tumour location necessitating an urgent therapeutic intervention (e.g., palliative care, surgery, or radiation therapy), such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture.
* Patients with progressive HNSCC within 6 months of completion of systemic therapy for locoregionally advanced disease with curative intent.
* Receiving treatment for brain metastases or leptomeningeal disease (LMD) which may interfere with safety and/or endpoint assessment. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to trial entry, have discontinued corticosteroid treatment for these metastases and are clinically stable, off anticonvulsants for at least 4 weeks and are neurologically stable before enrollment.
* Patients for whom single agent pembrolizumab is not the preferred treatment (e.g. patients for whom chemotherapy or anti-PD-1 in combination with chemotherapy is considered the preferred therapy by the investigator or treating physician).
* Prior treatment with any anti signal regulatory protein alpha (SIRPα) or anti-integrin-associated protein (CD47) agent, regardless of treatment intent.
* Prior cancer treatment with any anti PD-1 or anti PD-L1 agent or with an agent directed to another stimulatory or co-inhibitory Tcell receptor (e.g. CTLA-4, OX 40, CD137), regardless of treatment intent.
* Prior allogeneic stem cell or solid organ transplantation.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response (OR) with confirmation | Up to 27 months
  OR defined as the best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to response evaluation criteria in solid tumours version 1.1 (RECIST v1.1).
  Objective response (OR) will be defined by investigator's assessment from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, lost to follow-up or withdrawal of consent.

SECONDARY OUTCOMES:
Occurrence of treatment related adverse event (AE) from first treatment administration until the earliest of 90 days after the last dose, death, subsequent anti-cancer therapy, lost to follow-up or withdrawal of consent | Up to 27 months
Occurrence of treatment related AE leading to treatment discontinuation from first treatment administration until the earliest of 90 days after the last dose, death, subsequent anti-cancer therapy, lost to follow-up or withdrawal of consent | Up to 27 months
Overall survival (OS) | Up to 27 months
  OS defined as the time from first treatment administration until death from any cause.
Overall survival at 6 and 12 months (OS6 and OS12) | At 6 months and 12 months
  OS defined as being alive at 6 months or at 12 months from first treatment administration.
Progression-free survival (PFS) | Up to 27 months
  PFS defined as the time from first treatment administration until disease progression (PD) according to RECIST v1.1 or death from any cause, whichever occurs earlier.
Progression-free survival at 6 months (PFS6) | At 6 months
  PFS defined as being alive and without progression at 6 months from first treatment administration.
Duration of objective response (DOR) | Up to 27 months
  DOR defined as the time from first documented CR or PR (RECIST v1.1) until the earliest of PD or death among patients with OR.

CONTACTS AND LOCATIONS:
Locations (59):
- United States (3):
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - M Health Fairview Clinics and Surgery Center - Minneapolis, Minneapolis, Minnesota
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
- Australia (2):
  - Gosford Hospital, Gosford, New South Wales
  - Andrew Love Cancer Centre, Geelong, Victoria
- Brazil (3):
  - Hospital de Amor, Barretos
  - Liga Norte Riograndense contra o cancer, Natal
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
- MBAL Sveta Sofia, Sofia, Bulgaria
- France (4):
  - CTR Oscar Lambret, Lille
  - CTR Leon Berard, Lyon
  - HOP Timone, Marseille
  - INS Gustave Roussy, Villejuif
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- Germany (4):
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitätsklinikum Jena, Jena
  - Universität Leipzig, Leipzig
  - Universitätsklinikum Ulm, Ulm
- Hungary (3):
  - Semmelweis University, Budapest
  - National Institute of Oncology, Budapest
  - Clinexpert Gyongyos, Gyöngyös
- Italy (5):
  - Istituto Scientifico Romagnolo, Meldola (FC)
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Istittuo Nazionale Tumori Regina Elena - IRCCS, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (5):
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Kobe University Hospital, Hyogo, Kobe
  - Kansai Medical University Hospital, Osaka, Hirakata
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- Mexico (3):
  - Unidad Clinica Farmacologica Bioemagno, Mexico City
  - Instituto Nacional de Cancerologia, México
  - Centro Oncológico Internacional, Tlajomulco de Zuñiga
- ARENSIA Exploratory Medicine, Chisinau, Moldova
- Poland (2):
  - National Oncology Institute Maria Sklodowskiej Curie State Research Institute, Gliwice
  - Center of Oncology of the Lublin Region St. Jana z Dukli, Lublin
- "Prof. Dr. Alexandru Trestioreanu" Oncology Institut, Bucharest, Romania
- National University Hospital-Singapore-22806, Singapore, Singapore
- South Korea (3):
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, St.Vincent's Hospital, Suwon
- Spain (3):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (2):
  - Cantonspital Aarau, Aarau
  - University Hospital Zurich, Zurich
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Siriraj Hospital, Bangkoknoi, Thailand
- Turkey (Türkiye) (6):
  - Adana City Hospital, Adana
  - Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Hacettepe University Oncology Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Istanbul University Medical Faculty Capa Hospital, Istanbul
  - Ege University Tulay Aktas Oncology Hospital, Izmir
- United Kingdom (3):
  - St Bartholomew's Hospital, London
  - The Royal Marsden Hospital, Chelsea, London
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com